CLINICAL TRIAL: NCT03072381
Title: The Clinical, Biomechanical, and Tissue Regenerating Effects of a Single PEAK Platelet Rich Plasma Injection for the Treatment of Chronic Lateral Epicondylosis: a Randomized Controlled Trial
Brief Title: PEAK Platelet Rich Plasma Injection Treatment for Chronic Lateral Epicondylosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-0086; A536110 (Other: UW Madison); SMPH\ORTHOPEDIC&REHAB\ORTHO (Other: UW Madison); Protocol Version 3/10/2017 (Other: UW Madison)
Record Dates: First submitted 2016-11-08; First posted 2017-03-07 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Chronic Lateral Epicondylosis
Keywords: CLE; epicondylosis; platelet rich plasma; PRP; ultrasound; shear wave ultrasound; tendinopathy; elbow; tenis elbow; plasma; plasma injection; tendinosis; tendinitis
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma - Group 1 (Active Comparator): Subjects in Group 1 (PRP) will receive a single ultrasound-guided intratendinous (common extensor tendon origin) injection of up to 3 mL autologous PEAK platelet-rich plasma at week 0 (baseline).
  If a subject has bilateral elbow common extensor tendon pain, both elbows will be treated in the same study arm.
  Interventions: Biological: Platelet Rich Plasma - Group 1
- Corticosteroid Control - Group 2 (Placebo Comparator): Subjects in Group 2 (corticosteroid control) will receive a single ultrasound-guided intratendinous injection approximately (may be limited by tendon/soft tissue limitations of the subject) of 2 mL 1% lidocaine + 1mL of him 40mg Kenalog (triamcinolone hexacetonide, 40mg/mL) at week 0.
  If a subject has bilateral elbow common extensor tendon pain, both elbows will be treated in the same study arm.
  Interventions: Drug: Corticosteroid Control - Group 2

INTERVENTIONS:
Biological: Platelet Rich Plasma - Group 1 — Subjects in Group 1 (PRP) will receive a single ultrasound-guided intratendinous (common extensor tendon origin) injection of up to 3 mL autologous PEAK platelet-rich plasma at week 0 (baseline).
  Arms: Platelet Rich Plasma - Group 1
Drug: Corticosteroid Control - Group 2 — Subjects in Group 2 (corticosteroid control) will receive a single ultrasound-guided intratendinous injection approximately (may be limited by tendon/soft tissue limitations of the subject) of 2 mL 1% lidocaine + 1mL of him 40mg Kenalog (triamcinolone hexacetonide, 40mg/mL) at week 0.
  Arms: Corticosteroid Control - Group 2

SUMMARY:
The proposed project will be the first to assess pain- and function-dependent, elbow-specific quality of life and in-vivo mechanical properties of common extensor tendons post-treatment with PRP in a Level 1, RCT with subject and assessor blinding. The valuable data gained will significantly add to the knowledge base of treatment effects of PRP for a chronic tendinopathy. Positive findings of PRP compared to control (corticosteroid injection) would suggest future larger scale studies to help establish an optimal protocol for the nonsurgical management of CLE. Correlating US and shear wave acoustoelastography imaging assessments with validated clinical outcomes will provide a powerful tool for future outcomes analyses using a non-invasive imaging modality to monitor tissue healing both morphologically as well as biomechanically, and may even be used to evaluate injury risk.

DETAILED DESCRIPTION:
Randomization procedures Subjects will be randomized to 1 of 2 study arms. Subjects in Group 1 (PRP) will receive a single ultrasound-guided intratendinous (common extensor tendon origin) injection of up to 3 mL autologous PEAK platelet-rich plasma at week 0 (baseline). Subjects in Group 2 (corticosteroid control) will receive a single ultrasound-guided intratendinous injection approximately (may be limited by tendon/soft tissue limitations of the subject) of 2 mL 1% lidocaine + 1mL of him 40mg Kenalog (triamcinolone hexacetonide, 40mg/mL) at week 0. If a subject has bilateral elbow common extensor tendon pain, both elbows will be treated in the same study arm.

Blinding: Subjects and assessors will be blinded to the subject group allocation. Control subjects will also undergo phlebotomy to maintain blinding. Injection syringes will be cloaked using opaque adhesive tape in order to ensure the injector is unaware of subject treatment allocation. Subjects will be identified to study personnel using a unique study number only and results of the imaging studies will be blinded, batched and evaluated in a randomized manner.

Ultrasound imaging analyses will be conducted at baseline, 26 weeks, and 52 weeks post treatment.

The platelet concentration will be analyzed in both samples (whole blood compared to PRP) in order to record and verify the consistency of the concentration factor in PRP.

Shear wave ultrasound imaging will be compared using comparison of average shear wave speed (SWS) between baseline and post treatment 52 week follow-up between the two randomized groups. Shear wave speed is a quantitative measure obtained by measuring speed of ultrasound in a selected region of interest (ROI). In prior studies, the study team has successfully blinded the investigator when selecting the ROI, and conducted inter-rater repeatability analysis showing that this was a valid, repeatable way of measuring SWS in a particular ROI.

For patients:Total of 9 visits Initial Screen - Initial Eligibility Screening Baseline - Informational Meeting: Secondary eligibility screen, enrollment (informed consent), questionnaires; Grip Strength Test; Ultrasound and SWAE imaging Week 0 Intervention - Injection of PRP under ultrasound Weeks 4, 8, 12, 16 - Questionnaires: QUICK-DASH, SF-12, PRTEE, SANE-ELBOW, PRP Satisfaction; Grip Strength Test Week 26 - Questionnaires: QUICK-DASH, SF-12, PRTEE, SANE-ELBOW, PRP Satisfaction; Grip Strength Test; Ultrasound and SWAE imaging Week 52 - Questionnaires: QUICK-DASH, SF-12, PRTEE, SANE-ELBOW, PRP Satisfaction; Grip Strength Test; Ultrasound and SWAE imaging

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65
2. chronic (>3months) unilateral or bilateral common extensor tendon pain
3. clinical exam findings consistent with CLE
4. imaging confirmation of CLE (U/S or MRI)
5. self-reported failure of supervised physical therapy; 6) self-reported failure of at least 2 of the most common treatments (NSAIDs, relative rest, ice, bracing) for CLE.

Exclusion Criteria:

1. inability to comply with follow-up requirements of study
2. history of bleeding disorders, low-platelet counts, other hematologic conditions
3. elbow pain with other possible etiologies (e.g., degenerative joint disease)
4. currently using anticoagulation or immunosuppressive therapy
5. anticoagulant or immunosuppressive therapy within the prior month
6. known allergy to Lidocaine
7. self-reported pregnancy
8. worker's compensation injury
9. pending litigation
10. concurrent opioid use for pain
11. corticosteroid injection within the past 3 months
12. minors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Change in the QUICK-DASH upper limb disability questionnaire | one year (52 weeks)
  Patients receiving a single PRP PEAK injection for CLE will report improved Quick-DASH upper limb disability questionnaire from baseline to 52 week follow-up compared to control subjects (corticosteroid group)

SECONDARY OUTCOMES:
Ultrasound evaluation of changes of pathologic features | one year (52 weeks)
  Improved ultrasound (US) changes of several pathologic features of CLE as evaluated using US imaging of the common extensor tendon from baseline to 52 weeks post-treatment compared to control subjects. Conventional ultrasound will be done to assess thickness (contralateral comparison), neovascularity, and hypoechogenicity; and Acoustoelastography (AE) will be done to measure stiffness changes of the patellar tendon using standardized 0-3 severity scales compared to control subjects.

OTHER OUTCOMES:
Evaluation of subject satisfaction of PRP therapy | one year (52 weeks)
  Outcome measures will be compared for satisfaction with PRP therapy as assessed by the treatment satisfaction survey score at 52 weeks post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John J. Wilson, MD, MS, Principal Investigator — University of Wisconsin-Madison School of Medicine & Public Health
Locations (1):
- Wisconsin Institute of Medical Research (WIMR), Madison, Wisconsin, United States

REFERENCES:
- [Derived] Karjalainen TV, Silagy M, O'Bryan E, Johnston RV, Cyril S, Buchbinder R. Autologous blood and platelet-rich plasma injection therapy for lateral elbow pain. Cochrane Database Syst Rev. 2021 Sep 30;9(9):CD010951. doi: 10.1002/14651858.CD010951.pub2. PMID 34590307